CLINICAL TRIAL: NCT02311595
Title: A Phase II Clinical Trial of Reduced Port Totally Laparoscopic Distal Gastrectomy With D2 Lymph Node Dissection for Gastric Cancer Patients
Brief Title: A Phase II Clinical Trial of Reduced Port Totally Laparoscopic Distal Gastrectomy With D2 Lymph Node Dissection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-10-032
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; laparoscope
MeSH Terms: conditions — Stomach Neoplasms

ARMS (1):
- reduced port (Experimental): gastric cancer patients go through reduced port laparoscopic distal gastrectomy with D2 lymph node dissection
  Interventions: Procedure: reduced port laparoscopic distal gastrectomy

INTERVENTIONS:
Procedure: reduced port laparoscopic distal gastrectomy

SUMMARY:
The purpose of this study is to determine if reduced port totally laparoscopic distal gastrectomy with complete D2 lymph node dissection for gastric cancer is safe and oncological feasible.

67 patients with gastric cancer with preoperative staging from T1 to T3 will undergo reduced port totally laparoscopic distal gastrectomy.

The primary end point of this study is to measure compliance rate with pathology report and compare with previous compliance rate data.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the stomach
* Eastern Cooperative Oncology Group Eastern Cooperative Oncology Group performance status 0-1,
* signed informed consent
* location of the primary tumor in the antrum, angle and lower body
* no evidence of distant metastasis or invasion to adjacent organs or serosal infiltration

Exclusion Criteria:

* metastatic disease
* previous history of malignancy in any organ
* any co-morbidity obviating major surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Compliance rate (Japanese Research Society of Gastric Cancer (JRSGC) lymph node grouping) | 1 month after enrollment of the patients
  Compliance rate : Cases with no more than one missing lymph node station according to the Japanese Research Society of Gastric Cancer (JRSGC) lymph node grouping

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ho Lee, M.D. ph.D, Study Chair — Samsung Medical Center

REFERENCES:
- [Background] Lee JH, Kim YW, Ryu KW, Lee JR, Kim CG, Choi IJ, Kook MC, Nam BH, Bae JM. A phase-II clinical trial of laparoscopy-assisted distal gastrectomy with D2 lymph node dissection for gastric cancer patients. Ann Surg Oncol. 2007 Nov;14(11):3148-53. doi: 10.1245/s10434-007-9446-0. Epub 2007 Aug 20. PMID 17705092
- [Background] Kim SM, Lee JH, Lee SH, Ha MH, Seo JE, Kim JE, Choi MG, Sohn TS, Bae JM, Kim S. Techniques of reduced PRT laparoscopy-assisted distal gastrectomy (duet LADG). Ann Surg Oncol. 2015 Mar;22(3):793. doi: 10.1245/s10434-014-4087-6. Epub 2014 Sep 17. PMID 25227307
- [Background] Bonenkamp JJ, Hermans J, Sasako M, van de Velde CJ, Welvaart K, Songun I, Meyer S, Plukker JT, Van Elk P, Obertop H, Gouma DJ, van Lanschot JJ, Taat CW, de Graaf PW, von Meyenfeldt MF, Tilanus H; Dutch Gastric Cancer Group. Extended lymph-node dissection for gastric cancer. N Engl J Med. 1999 Mar 25;340(12):908-14. doi: 10.1056/NEJM199903253401202. PMID 10089184